CLINICAL TRIAL: NCT01435057
Title: Monocentric, Randomized, Controlled Study for Reduction on Visceral Fat Dynamic and Resting Energy Expenditure in Obese Patients Via Strength Versus Endurance Training (STEN Study - STrength Versus ENdurance Training)
Brief Title: Effects of Different Exercise Training Regimens on Visceral Fat Dynamic and Resting Energy Expenditure in Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Matthias Bluher, medical doctor, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEN
Record Dates: First submitted 2011-05-11; First posted 2011-09-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Abdominal Obesity
Keywords: Abdominal Obesity; training; fat; insulin; glucose; diet
MeSH Terms: conditions — Obesity, Abdominal; Platelet Glycoprotein IV Deficiency; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endurance training (Active Comparator): Endurance training:
  Supervised, twice a week, each training session consists of a 20 min warm up and cool down period and a minimum of 40min tread mill, rawing device or bicycle training.
  During the study period of 24 months, we will perform an open randomized, prospective training intervention study comparing the effects of three times a week either strength or endurance training on reduction of visceral fat area as determined by MRI scans at the level of L4-L5.
  Interventions: Procedure: exercise training
- strength training (Active Comparator): Strength training:
  Supervised, twice a week, each training session consists of a 20 min warm up and cool down period and a minimum of 40min circle training
  During the study period of 24 months, we will perform an open randomized, prospective training intervention study comparing the effects of two to three times a week either strength or endurance training on reduction of visceral fat area as determined by MRI scans at the level of L4-L5.
  Interventions: Procedure: exercise training

INTERVENTIONS:
Procedure: exercise training — comparison of strength versus endurance training (two or three times a week, 60 minutes per training session) over 24 months

SUMMARY:
In this project, the investigators will test the hypothesis that predominant (two to three times a week 60 min) strength training is more effective in reducing visceral fat mass than endurance training in obese patients.

DETAILED DESCRIPTION:
Strength training (ST) was shown to be more effective than endurance training (ET) in improving glycemic control in the treatment of type 2 diabetes. However, it is unknown, whether different training strategies have different effects on the preferential visceral adipose tissue reduction and changes in resting energy expenditure in a population with abdominal obesity. We will therefore compare ST and ET (two to three times a week, 60 minutes per training session) in addition to a restricted energy intake of 1500kcal per day for women and 1800kcal per day for men in a prospective study of 200 individuals with abdominal obesity defined by a waist circumference > 102 cm for males and > 88 cm for females and a BMI > 35 kg/m² with regard to:

1. Abdominal visceral adipose tissue area dynamic (MRI studies)
2. Abdominal subcutaneous adipose tissue area dynamic (MRI studies)
3. Total body fat mass changes (bioelectrical impedance analysis)
4. Changes in resting energy expenditure (indirect calorimetry)
5. Changes in parameters of glucose metabolism, insulin sensitivity and lipid profile
6. Changes in circulating adipokines and markers of inflammation In addition, we will search for novel serum parameters, which predict the individual training response by a serum metabolomics/ proteomics approach.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 35 kg/m2
* waist circumference >102cm (men), >88cm (women)
* age 18 - 60 years
* written informed consent

Exclusion Criteria:

* type 1 or type 2 diabetes
* fasting plasma glucose >= 6.0 mmol/l
* 2h-OGTT (oral glucose tolerance test) glucose >= 11.1 mmol/l
* any chronic inflammatory or malignant disease
* medical treatment which influences glucose metabolism
* drug or alcohol abuse
* psychiatric disorders
* untreated thyroid dysfunction
* cardiac pacemaker or other contraindication for MRI
* attendant therapy with oral antidiabetic medication, GLP-1 mimetics or analoga, Insulin, anti-obesity medication (orlistat, sibutramine), Falithrom, antipsychotic drugs, any chemotherapeutics
* pregnant or nursing women
* expected low compliance
* current participation in another investigational trial
* last exercise training <= 6 months ago

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
MRI | Baseline and after 12 months after randomisation
  Change from Baseline in abdominal visceral fat area as determined by MRI scans at the level of L4-L5 after 12 months of training intervention

SECONDARY OUTCOMES:
MRI | Baseline, 12 and 24 months after randomisation
  Changes from Baseline in abdominal visceral and subcutaneous fat area
BIA | Baseline, 6, 12, 18 and 24 months after randomisation
  Changes from Baseline in total body fat mass
compliance to the intervention | over 24 months of intervention
  compliance to the intervention of training (strength or endurance) as measured by the number of realized training units. Non-compliance = cumulative time bigger than six weeks per year
well being as measured by SF-36 | Baseline and every 6 months during intervention
  Changes from Baseline in individual well being as measured by SF-36
indirect calorimetry | Baseline, 6, 12, 18 and 24 months after randomisation
  Changes from Baseline in resting energy expenditure
fasting plasma glucose | Baseline and every 12 months
  Changes from Baseline in fasting plasma glucose, insulin sensitivity and insulin secretion determined in oral glucose tolerance tests
inflammatory parameters | Baseline and every 3 months during intervention
  Changes from Baseline in inflammatory parameters
adipokine serum concentrations | Baseline and every 3 months during intervention
  Changes from Baseline in adipokine serum concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Blüher, prof., MD, Principal Investigator — University of Leipzig
Locations (1):
- University of Leipzig, Department of Medicine, Leipzig, Saxony, Germany